CLINICAL TRIAL: NCT07319234
Title: MENU: A Novel Family-Driven Approach to Support Families Awaiting Autism Diagnostic Evaluation
Brief Title: Development of MENU Protocol
Acronym: MENU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Baylor University (Other)
Responsible Party: Principal Investigator, James D Lee, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MENU study
Record Dates: First submitted 2025-11-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Autism; Mental Health
Keywords: autism; mental health; diagnostic evaluation waitlist
MeSH Terms: conditions — Autistic Disorder; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MENU group (Experimental): The group receive modular content drawn from three well-established practices targeting core characteristics of autism: Acceptance and Commitment Therapy for caregiver mental health and well-being, Enhanced Milieu Teaching for child social communication, and RUBI behavioral parent training for managing challenging behaviors.
  Interventions: Behavioral: MENU

INTERVENTIONS:
Behavioral: MENU — The intervention consists of modular content drawn from three well-established practices targeting core characteristics of autism: Acceptance and Commitment Therapy for caregiver mental health and well-being, Enhanced Milieu Teaching for child social communication, and RUBI behavioral parent training for managing challenging behaviors. In this model, caregivers work with the research team to select and sequence modules based on their needs, preferences, and priorities, making MENU highly personalized, family-centered, and accessible. Families will engage with MENU modules over 16 weeks, although exact duration may vary based on individual family goals and pacing.

SUMMARY:
The overarching goal of this project is to reduce autism-related health disparities. The investigators will develop and pilot MENU, a culturally responsive and caregiver-driven intervention specifically designed to support underserved families of young autistic children during the diagnostic wait period. MENU will equip underserved caregivers with flexible, evidence-based strategies to improve parent mental health, child social communication, and challenging behaviors. The intervention consists of modular content drawn from three well-established practices targeting core characteristics of autism: Acceptance and Commitment Therapy for caregiver mental health and well-being, Enhanced Milieu Teaching for child social communication, and RUBI Parent Training for managing a child's challenging behaviors.

In this model, caregivers collaborate with the research team to select and sequence modules based on individual needs, preferences, and priorities, making MENU highly personalized, family-centered, and accessible. Families will engage with MENU modules over approximately 12 weeks, with duration varying based on individual goals and pacing. The project utilizes a explanatory, sequential mixed methods design, an approach that examines preliminary effectiveness and gathers detailed information on contextual factors relevant to future scale-up and sustainability within public systems of care in Texas, including Part C Early Intervention programs. Up to 50 underserved families representing diverse racial, ethnic, and linguistic backgrounds will be recruited in strategic partnership with trusted community organizations throughout Texas. To maximize accessibility and reduce barriers associated with the digital divide, the project will provide iPads and cellular data plans to families lacking adequate Internet access or devices. Following comprehensive baseline assessments, including standardized measures and clinical interviews, caregivers will collaborate with the research team to select and tailor MENU modules aligned with individual goals and needs across the three evidence-based practices. Quantitative data will be collected at baseline, immediately post-intervention, and at 3-month follow-up using validated measures of parent mental health, child social communication, and challenging behaviors. Implementation outcomes (e.g., acceptability, feasibility, usability) will be assessed in partnership with community advisors, with regular reviews informing iterative refinements to maintain cultural and contextual relevance for Texas families. By pioneering scalable supports delivered before a formal autism diagnosis, MENU challenges conventional service timelines and introduces a new model of early autism care in Texas. The project will also generate actionable data to inform policy shifts, reimbursement pathways, and integration into early childhood systems, contributing to reductions in health and educational disparities among autistic children and their families.

DETAILED DESCRIPTION:
This project addresses health disparities by offering proactive support during a critical period when services are typically unavailable to minoritized families due to systemic delays, insurance restrictions, and limited access to care. Early autism intervention is considered a gold standard for promoting optimal child and family outcomes, yet many families remain underserved due to a lack of diagnosis. MENU aims to mitigate this disparity by providing preemptive intervention prior to formal diagnosis to improve caregiver mental health, reduce developmental delays, and enhance families' capacity to advocate for their children. The broader impact of this approach includes reducing downstream educational and health disparities, informing public insurance policy, and establishing a scalable framework for equitable early autism intervention. By introducing high-quality, scalable supports delivered before a formal diagnosis, MENU challenges conventional service timelines and establishes a new model of early autism care in Texas and other states. Key implementation challenges include recruitment and retention of underserved families and maintaining cultural and contextual relevance while providing timely support. These challenges will be mitigated through partnerships with trusted community-based organizations composed of caregivers, service providers, and autistic self-advocates.

To support successful implementation, the project includes collaborations with grassroots organizations serving caregivers of autistic children (e.g., Texas Parent to Parent, Autism Society of Texas), racially or economically minoritized families (e.g., VELA, La Puerta Waco, Compassion Waco). Project success will be measured through quantitative and qualitative data aligned with the Project Work Plan. Outcome metrics include reductions in caregiver stress (Parenting Stress Index-Short Form), improvements in child communication (Vineland Adaptive Behavior Scales or Social Communication Questionnaire), improvements in challenging behaviors (Behavior Assessment System for Children), module completion rates, caregiver satisfaction, and implementation outcomes such as feasibility (Feasibility of Intervention Measure), acceptability (Acceptability of Intervention Measure), and usability (Intervention Usability Scale). Data will be collected at baseline, post-intervention, and follow-up, along with semi-structured interviews to assess sustained impact. The intervention period will last approximately 16 weeks, allowing sufficient time for meaningful engagement, skill acquisition, and observable outcomes. The project team includes interdisciplinary faculty members from the University of Texas at Austin and Baylor University with extensive experience supporting underserved families of young autistic children and strong research-practice partnerships. Community partners, including Texas Early Childhood Intervention agencies and minority-serving advocacy organizations, will contribute to participant recruitment, intervention refinement, validation, and statewide dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of young children between the ages of 2 and 5 years who were referred for autism diagnostic evaluation but have not yet been received services
* Caregivers from underserved populations, including families from racial and ethnic minority backgrounds (e.g., Latino and Black communities), rural communities, immigrant families, and Medicaid-eligible families in Texas
* Caregivers aged 18 years or older

Exclusion Criteria:

* Caregivers of children who have no concerns related to autism spectrum disorder
* Caregivers who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Adaptive Behavior Assessment System - Third Edition | Baseline (Day 1), immediately post-intervention (Week 12), and 1-month post-intervention follow-up (Week 16)
  Children's adaptive communication skills as measured by the Adaptive Behavior Assessment System, Third Edition (ABAS-3) Communication Domain. The Communication Domain consists of 26 items assessing receptive, expressive, and pragmatic communication skills in everyday contexts. Domain scaled scores range from 1 to 19, with higher scores indicating better adaptive communication functioning.
Patient Health Questionnaire - 8 | Baseline (Day 1), immediately post-intervention (Week 12), and 1-month post-intervention follow-up (Week 16)
  Caregiver depressive symptom severity as measured by the Patient Health Questionnaire-8 (PHQ-8), an 8-item self-report measure assessing the frequency of depressive symptoms over the past two weeks. Total scores range from 0 to 24, with higher scores indicating greater depressive symptom severity.
General Anxiety Disorder - 7 | Baseline (Day 1), immediately post-intervention (Week 12), and 1-month post-intervention follow-up (Week 16)
  Caregiver anxiety symptom severity as measured by the Generalized Anxiety Disorder 7-Item Scale (GAD-7), a 7-item self-report measure assessing the frequency of anxiety symptoms over the past two weeks. Total scores range from 0 to 21, with higher scores indicating greater anxiety symptom severity.
Home Situations Questionnaire - Autism Spectrum Disorder | Baseline (Day 1), immediately post-intervention (Week 12), and 1-month post-intervention follow-up (Week 16)
  Child disruptive behavior in everyday home situations as measured by the Home Situations Questionnaire-Autism Spectrum Disorder (HSQ-ASD). The HSQ-ASD is a caregiver-reported measure consisting of items assessing the severity of noncompliant and disruptive behaviors across common home situations. Total scores range from 0 to 9, with higher scores indicating greater severity of disruptive behavior.
caregiver satisfaction | immediately post-intervention (Week 12)
  a research-developed questionnaire to measure the caregiver's satisfaction of the intervention. It will be a 5 point Likert scale.
Feasibility of Intervention Measure | immediately post-intervention (Week 12)
  caregivers' rating of the feasibility of the implementation on a 5-point Likert scale
Acceptability of Intervention Measure | immediately post-intervention (Week 12)
  caregivers' acceptability of the intervention
Intervention Usability Scale | immediately post-intervention (Week 12)
  caregivers' rating of the usability of the intervention

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of concerns regarding participant privacy, limited resources for data sharing infrastructure